| Cover page: |
|---|
| Title: |
| Breathing Exercise for Chronic Pain Management in Breast Cancer Survivors: A Preliminary Randomized Controlled Trial |
| NCT 05257876 |
| 01/02/2023 |
| Informed consent: |

# **Charles Darwin University**

## College of Nursing and Midwifery

### Informed Consent Form (Draft version)

Breathing Exercise for Chronic Pain Management in Breast Cancer Survivors: A Preliminary
Randomized Controlled Trial

Student Investigator: Haiying Wang, PhD student, College of Nursing & Midwifery, Charles Darwin University, Australia

**Principal Investigator**: Professor Benjamin Tan, PhD, RN, College of Nursing & Midwifery, Charles Darwin University, Australia

#### Participant's declaration:

- I have read the Participant Information Sheet and fully understand the aims, objectives, and procedures of this study.
- ✓ I consent to participate in this pilot randomized controlled trial and the semi-structured interview which will explore my experience of participating in this pilot trial.
- I understand that I can ask any questions about this study and my questions will be answered properly by the researchers.
- ✓ I know that I will not receive any payment for participating in this study.
- ✓ I am voluntarily participating in this study, and I know that I have the full right to withdraw from the study at any time, which will not result in any negative consequences for me.
- I understand that if I withdraw from the study, the information I provided will not be used for this study.
- I understand that the researchers will keep my personal information confidential so far as the law allows
- I understand that the information obtained from this research will be used in future research and published in academical journals or presented at conferences, but my right to privacy will be retained.

Date:

- ✓ I agree that all the data collected from the study will only be used for scientific study.
- ✓ I agree to be contacted by phone call.
- ✓ I agree to be audio-recorded during the semi-structured interview.
- ✓ I agree to receive video calls as necessary.

#### I have read, understand, and agree with all the terms in this consent form.

| I have explained the aims, objectives, proceed participant and answered all questions, and explanation. | |
|---|---|
| Researcher's name: | |
| Researcher's signature: | Date: |

COLLEGE OF

Participant's name:

Participant's signature:

Researcher's declaration:

NURSING AND MIDWIFERY

ALICE SPRINGS BRISBANE DARWIN MELBOURNE PERTH SYDNEY

CDU Casuarina Campus, Ellengowan Drive, Brinkin, Northern Territory, Australia 0811. CRICOS Provider No. 00300K (NT/VIC) | 03286A (NSW) KTD Provider No. 0373 | ABN 54 093 513 649 CHARLES
DARWIN
UNIVERSITY
AUSTRALIA